CLINICAL TRIAL: NCT04554550
Title: Post-operative Cognitive Function Following Pelvic Floor Surgery
Status: Completed | Type: Observational
Sponsor: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Uduak Andy, Assistant Professor of Obstetrics and Gynecology, University of Pennsylvania
Other Study IDs: 843178
Record Dates: First submitted 2020-09-12; First posted 2020-09-18 (Actual); Last update posted 2022-07-25 (Actual); Status verified 2022-07

CONDITIONS: Pelvic Organ Prolapse
MeSH Terms: conditions — Pelvic Organ Prolapse

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study is to assess cognitive function before and after surgery for pelvic organ prolapse using sensitive tests of various neurocognitive domains.

DETAILED DESCRIPTION:
Post operative cognitive dysfunction has been well described as a relatively common phenomenon with potentially long-lasting detrimental effects. However, there are currently limited data exploring the effects of gynecologic surgery on cognitive function. The population of patients treated surgically for pelvic floor disorders is typically older, and therefore at higher baseline risk for cognitive dysfunction. Therefore, it is of interest to determine the effects of pelvic floor surgery and anesthesia on this patient population. The investigators plan to conduct a prospective cohort study to assess cognitive function before and after pelvic organ prolapse surgery using sensitive tests of memory and other neurocognitive domains. Participants will be women undergoing surgery for pelvic organ prolapse. All participants will undergo cognitive tests at three time points: at their pre-operative clinic appointment, in the hospital the morning after surgery, and at their post-operative clinic appointment. In addition to the neurocognitive tests, patients will undergo a series of questionnaires regarding physical function, frailty, sleep quality, and incontinence symptoms.

ELIGIBILITY:
Inclusion Criteria: Women 60 years of age or older who are scheduled to undergo surgery for pelvic organ prolapse.

Exclusion Criteria:

* Women who have a known baseline diagnosis of cognitive dysfunction or central nervous disorder
* A Mini-Mental State Exam (MMSE) score of greater than 24
* Non-english speaking
* Any severe visual or auditory disorder
* Alcoholism or drug dependence

Min Age: 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women aged 60 and older scheduled to undergo surgery for pelvic organ prolapse at the University of Pennsylvania.
Sampling Method: Non-Probability Sample
Enrollment: 130 (Actual)
Dates: Start 2020-08-13 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
Change in episodic memory neurocognitive test scores | 8 weeks
  Episodic memory will be assessed using the Scene Encoding/Recognition Test

CONTACTS AND LOCATIONS:
Overall Officials: Uduak Andy, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No